CLINICAL TRIAL: NCT06752798
Title: Bone Marrow Protective Effect of Trilaciclib in Postoperative Concurrent Chemoradiotherapy for Locally Advanced Head and Neck Squamous Cell Carcinoma: An Open-Label, Single-Arm, Phase 2 Clinical Study
Brief Title: Bone Marrow Protective Effect of Trilaciclib in Postoperative CCRT for LA-HNSCC
Acronym: CCRT，LA-HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-HNSCC-001
Record Dates: First submitted 2024-12-07; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Cancer Squamous Cell Carcinoma
Keywords: Trilaciclib; Head and neck cancer; Adjuvant treatment; chemoradiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — trilaciclib; Cisplatin

STUDY DESIGN:
Intervention Model Description: Single-group assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trilaciclib + Cisplatin (Experimental): Trilaciclib: 240 mg/m², intravenous infusion over 30 minutes, administered within 4 hours prior to each chemotherapy session.
  Cisplatin: 40 mg/m², intravenous infusion over 2-3 hours, once a week, for a total of 6-7 times.
  Interventions: Drug: Trilaciclib + Cisplatin

INTERVENTIONS:
Drug: Trilaciclib + Cisplatin — Trilaciclib: 240 mg/m², intravenous infusion over 30 minutes, administered within 4 hours prior to each chemotherapy session. Cisplatin: 40 mg/m², intravenous infusion over 2-3 hours, once a week, for a total of 6-7 times.

SUMMARY:
To evaluate the efficacy and safety of trilaciclib combined with standard treatment project as an adjuvant treatment for Head and neck cancer after surgery

DETAILED DESCRIPTION:
Trilaciclib indication: Trilaciclib, a CDK4/6 inhibitor, was used before chemotherapy to reduce the incidence of bone marrow suppression and approved by the FDA for small cell lung cancer patients in 2021.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be enrolled in this study:

  * Pathologically or histologically confirmed locally advanced squamous cell carcinoma of the head and neck (this study includes cancers of the oral cavity, oropharynx, hypopharynx, and larynx, excluding cancers of the lip and nasopharynx).
  * Indications for surgery and postoperative chemotherapy plus radiotherapy, and meeting the following conditions:
* (1) Staging of T1-4N0-3M0, having undergone radical surgery;
* (2) At least one of the following factors: positive surgical margin, tumor close to the surgical margin, postoperative pathological staging pT3-4 or pN2-3, positive lymph nodes in neck level IV or V, tumor invasion of nerves/blood vessels/lymphatic vessels.

  * ECOG performance status score of 0-1.
  * Normal major organ function, meeting the following criteria:
* (1) Hematology standards (no blood transfusion or blood products within 14 days): a. HB ≥ 90 g/L; b. Neu ≥ 1.5×10^9/L; c. PLT ≥ 100×10^9/L;
* (2) Biochemical criteria: a. TBIL < 1.5× upper limit of normal (ULN); b. ALT and AST < 2.5× ULN; c. Serum Cr ≤ 1.0× ULN or creatinine clearance rate > 60 ml/min.

  * Women of childbearing potential must have a negative pregnancy test (serum or urine) within 7 days prior to enrollment and must agree to use reliable contraception during the study and for a specified period after the last dose of the study drug.
  * Women of childbearing potential must have taken reliable contraceptive measures or have a negative pregnancy test (serum or urine) within 7 days prior to enrollment, and must agree to use appropriate contraceptive methods during the study and for 8 weeks after the last dose of the study drug. For male participants, they must agree to use appropriate contraceptive methods during the study and for 8 weeks after the last dose of the study drug or have undergone surgical sterilization.
  * The subjects voluntarily join this study and sign the informed consent form.

Exclusion Criteria:

* Pathologically confirmed non-squamous cell carcinoma.
* Patients with recurrence or distant metastasis (M1).
* Previous chemotherapy for any reason, or prior surgery, radiotherapy, molecular targeted therapy, or immune checkpoint inhibitor therapy (anti-PD-1, anti-PD-L1, anti-PD-L2, etc.) in the head and neck region.
* Pregnant or breastfeeding women.
* Previous or concurrent other malignancies.
* Patients with other uncontrolled serious diseases.
* Abnormal function of vital organs such as the heart, brain, or lungs: Hypertension that cannot be controlled to normal range with antihypertensive drugs (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90mmHg); Grade I or higher myocardial ischemia or myocardial infarction, arrhythmia, and Grade II heart failure; stroke or cardiovascular events within 6 months prior to enrollment; abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with a tendency to bleed or receiving thrombolytic or anticoagulant therapy; clear tendency to bleed; patients with positive proteinuria (urine protein test 2+ or above, or 24-hour urine protein quantification > 1.0 g).
* Active infections requiring systemic treatment, such as tuberculosis.
* Previous hematopoietic stem cell or bone marrow transplant.
* Known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1/2 antibody positive).
* Untreated active hepatitis B; Note: Hepatitis B subjects meeting the following criteria are eligible: HBV viral load must be < 1000 copies/ml (200 IU/ml) before the first dose, and subjects should receive anti-HBV therapy throughout the study chemotherapy to prevent viral reactivation. For subjects who are anti-HBc (+), HBsAg (-), anti-HBs (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring for viral reactivation is necessary; active HCV infection subjects (HCV antibody positive and HCV-RNA levels above the detection limit).
* History of substance abuse that cannot be abstained from or mental disorders.
* Allergy to the study drug or its components.
* Any other conditions that the investigator judges may affect the conduct of the clinical study and the determination of the study results.
* Concurrent participation in another therapeutic clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade 3/4 Neutropenia | From the date of enrollment to the 15th day after the completion of postoperative concurrent chemoradiotherapy.
  Neutrophils ≤ 1.0*109/L

SECONDARY OUTCOMES:
Incidence of Grade 3/4 Thrombocytopenia during Chemotherapy | From the date of enrollment to the 15th day after the completion of postoperative concurrent chemoradiotherapy.
  Platelets≤ 50*109/L
Incidence of Grade 3/4 Anemia during Chemotherapy | From the date of enrollment to the 15th day after the completion of postoperative concurrent chemoradiotherapy.
  hemoglobin<80g/L
Incidence of Febrile Neutropenia | From the date of enrollment to the 15th day after the completion of postoperative concurrent chemoradiotherapy.
  ANC <0.5×10^9/L or ANC between 0.5 and 1×10^9/L (Grade 3) but expected to drop to <0.5×10^9/L within the next 48 hours;temperature ≥38.3°C or ≥38.0°C for more than 1 hour.
Incidence of Platelet Transfusion | From the date of enrollment to the 15th day after the completion of postoperative concurrent chemoradiotherapy.
  Incidence of Platelet Transfusion
Incidence of Red Blood Cell Transfusion | From the date of enrollment to the 15th day after the completion of postoperative concurrent chemoradiotherapy.
  Incidence of Red Blood Cell Transfusion

OTHER OUTCOMES:
Survival Data-Related Endpoints | 1-Year
  1-Year Disease-Free Survival (DFS) Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes